CLINICAL TRIAL: NCT06272279
Title: Neuromodulation With Spinal Stimulation Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS23666(B2020:015)
Record Dates: First submitted 2021-03-09; First posted 2024-02-22 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury at C5-C7 Level; Paraplegia, Spinal; Paraplegia, Incomplete
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Intervention Model Description: Semi-blinded, randomized block entry design, crossover intervention study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be connected to the stimulation device(s) but will not know if it has been turned on during each trial. In addition, the person analyzing the outcome data will not be aware of the stimulation status of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal cord stimulation (Experimental): Spinal cord stimulation will be administered to participants for 15 min.
  Interventions: Device: spinal stimulation-DCS; Other: spinal stimulation-EPS
- Shamspinal cord stimulation (Sham Comparator): Sham spinal cord stimulation will be administered to participants for 15 min.
  Interventions: Other: spinal stimulation-sham DCS; Other: sham spinal stimulation-EPS

INTERVENTIONS:
Device: spinal stimulation-DCS — transcutaneous spinal stimulation by direct current stimulation
  Arms: Spinal cord stimulation
Other: spinal stimulation-sham DCS — sham transcutaneous spinal stimulation by direct current stimulation
  Arms: Shamspinal cord stimulation
Other: spinal stimulation-EPS — transcutaneous spinal stimulation by electrical pulsed stimulation
  Arms: Spinal cord stimulation
Other: sham spinal stimulation-EPS — sham transcutaneous spinal stimulation by electrical pulsed stimulation
  Arms: Shamspinal cord stimulation

SUMMARY:
This is a pilot research study to test the protocols needed for transcutaneous spinal electrical stimulation in persons living with spinal cord injury (SCI). Up to 24 participants will be enrolled. A variety of stimulation parameters and outcome measures will be assessed.

DETAILED DESCRIPTION:
Purpose of this project

Spinal cord stimulation has the potential to improve motor function recovery after spinal cord injury. Commonly used approaches include low-intensity, direct current (DC) stimulation applied across multiple segments, electrical transcutaneous (ETC) stimulation, and magnetic transcutaneous stimulation (MTC).

Objective: to evaluate and compare the voluntary and reflexive motor performance in the same subjects, including people with and without spinal cord injury, after non-invasive spinal cord stimulation interventions. Comparing two different interventions applied in different experimental sessions and the respective sham stimulation is the goal of this study.

corticospinal and spinal motor pathways in paraplegics and in non-injured humans will be tested.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury C4 to L4
* ability to understand and follow directions

Exclusion Criteria:

* history of seizures, head injury, concussion, unexplained loss of consciousness or if they lived with an implanted cochlear stimulator, brain/neurostimulator, cardiac pacemaker, medication infusion device or live with metal implants in their body or if they are pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Motor response | Immediately after stimulation (within 1-15 min)
  H-reflex input output curve
Motor evoked potentials | Immediately after stimulation (within 1-15 min)
  MEP input-output curve

SECONDARY OUTCOMES:
Blood pressure | During the procedure/stimulation and up to 15 min after stimulation.
  Measured (in arm) with inflatable cuff-automated, standard machine.
Perception of discomfort due to stimulation | During and after procedure/stimulation and up to 15 min after stimulation.
  self-reporting on a scale ( the higher, the more discomfort)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request, we will consider making anonymized data available for analysis by other researchers
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study completion (May 2022) for one year.
Access Criteria: Upon request